CLINICAL TRIAL: NCT07357688
Title: The Effect of Acupuncture Therapy on Cognitive Function in Post-COVID-19 Myalgic Encephalomyelitis/Chronic Fatigue Syndrome: A Study With Multimodal Magnetic Resonance Imaging
Brief Title: The Effect of Acupuncture Therapy on Cognitive Function in Post-COVID-19 Myalgic Encephalomyelitis/Chronic Fatigue Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xi Wu (Other)
Responsible Party: Sponsor-Investigator, Xi Wu, Professor, Chengdu University of Traditional Chinese Medicine
Organization: Chengdu University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025KL-111
Record Dates: First submitted 2026-01-01; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Myalgic Encephalomyelitis/Chronic Fatigue Syndrome
Keywords: Post-COVID-19; myalgic encephalomyelitis/chronic fatigue syndrome; hippocampus; cognitive function; neurochemical; functional connectivity; multimodal MRI; acupuncture
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: data analysts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Verum acupuncture group (VA) (Experimental): Acupoint with acupuncture treatment
  Interventions: Other: Acupuncture
- Sham acupuncture group (SA) (Sham Comparator): Non-acupoint with sham acupuncture treatment
  Interventions: Other: Sham acupuncture
- Waitlist control group (No Intervention): Acupoint with acupuncture treatment after 8-week waiting period

INTERVENTIONS:
Other: Acupuncture — Participants will be alternatively acupunctured on two set of acupoints . The first set of acupuncture points incudes Baihui (GV20), bilateral Shenmen (HT7), bilateral Neiguan (PC6), Qihai (CV6), Guanyuan (CV4), bilateral Zusanli (ST36), bilateral Sanyinjiao (SP6). The second set of acupoints consist of Sishenchong (EX-HN1), bilateral Ganshu (BL18), bilateral Pishu (BL20), bilateral Shenshu (BL23), bilateral Taixi (KI3).The treatment consists of 24 sessions of 30 minutes, given within eight weeks (three sessions per week). A set of acupoints is acupunctured each treatment session.
  Arms: Verum acupuncture group (VA)
Other: Sham acupuncture — Nonpenetrating acupuncture on non-acupoints will be performed using Park sham acupuncture device (0.25 mm in diameter and 40 mm in length, Hwatuo, Suzhou, China) for participants. Two sets of non-acupoints will be alternatively acupunctured. The first set of sham acupoints includes bilateral non-acupoint 1, bilateral non-acupoint 2, non-acupoint 3, non-acupoint 4, bilateral non-acupoint 5, bilateral non-acupoint 6. The second set consists of bilateral non-acupoint 7, bilateral non-acupoint 8, bilateral non-acupoint 9, bilateral non-acupoint 10. The treatment consists of 24 sessions of 30 minutes, given within eight weeks (three sessions per week). A set of non-acupoints will be acupunctured each treatment session.
  Arms: Sham acupuncture group (SA)

SUMMARY:
Background of study:

Myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS) is a common sequela after SARS-CoV-2 infection(COVID-19). Cognitive dysfunction is one of the most common debilitating symptoms in ME/CFS. Currently, standardized therapy for ME/CFS has not been established. Some treatments, such as cognitive behavioral therapy (CBT) and graded exercise therapy (GET), mainly exert effects on physical symptoms, whereas the influence on cognitive problems is not significant. Acupuncture is an important complementary and alternative therapy for ME/CFS. However, However, research focused on the impact of acupuncture on cognitive functions in ME/CFS is rare. Additionally, no study has evaluated the efficacy and mechanism of acupuncture treatment in improving cognitive functions for post-COVID-19 ME/CFS.

Objective of the study:

The first objective of this study is to assess the efficacy of acupuncture treatment in improving cognitive function for post-COVID-19 ME/CFS. The second objective is to explore whether acupuncture improves cognitive ability in patients with post-COVID-19 ME/CFS through modulating hippocampal connectivity and metabolites using multimodal magnetic resonance imaging(MRI).

Study design:

A prospective, three-armed, randomized controlled trial with resting-state functional MRI(rs-fMRI) and magnetic resonance spectroscopy(MRS). Adults with post-COVID-19 ME/CFS will be randomly assigned to acupuncture, sham acupuncture, or waitlist control group in a 1:1:1 ratio, receiving 8-week intervention or waiting. Cognitive functions and resting-state functional connectivity(RSFC) and the levels of metabolites for each hippocampus will be examined at baseline and 8th week.

Study population:

Patients fulfilling 2015 National Academy of Medicine (NAM) criteria for ME/CFS following COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old
* Fatigue occurred during or after initial recovery of COVID-19 confirmed by nasopharyngeal swab reverse transcription-polymerase chain reaction(RT-PCR) or antigen testing lasts for at least 6 months
* Fulfilling US National Academy of Medicine(NAM) criteria for ME/CFS
* Chinese native speaker
* Right handedness
* Voluntary to participate in the study and signing the informed consent form.

Exclusion Criteria:

* Persistent fatigue occurs prior to COVID-19
* Previous or current diagnosis of severe chronic diseases such as heart, kidney or liver failure, tumor
* Previous or current diagnosis of neurological or psychiatric disorder such as neurodegenerative disease, stroke, epilepsy, bipolar disorder, schizophrenia
* Previous or current diagnosis of endocrine or metabolic disease such as hypothyroidism, adrenocortical hypofunction, type 2 diabetes
* Previous or current diagnosis of autoimmune disease such as systemic lupus erythematosus, Sjögren's syndrome, rheumatoid arthritis
* Chronic infection or inflammatory disease such as acquired immune deficiency syndrome(AIDS), chronic hepatitis, irritable bowel syndrome
* Substance or alcohol abuse
* Obesity (Body Mass Index≥28)
* Long-term use of immunosuppressant or glucocorticoid
* Within one year after major surgery
* Metal or electronic device implants
* Claustrophobia
* Pregnancy or lactation
* Previous acupuncture treatment in the latest 3 months
* Participating in another clinical research within a month

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change of Symbol Digit Modality Test score from baseline to the end of 8 weeks | Baseline and 8 weeks
  Symbol Digit Modality Test assesses attention through measuring the number of correct responses within 90 seconds. The minimum score is 0, and the maximum score is 110. Higher score indicates better attention.

SECONDARY OUTCOMES:
Changes of Digit Span Test scores from baseline to the end of 8 weeks | Baseline and 8 weeks
  Digit Span Test consists of forward and backward subtests, that respectively assess attention and executive function through measuring the number of correct digit sequences. The minimum score is 0 , and the maximum scores are respectively 10 and 9 for forward and backward subtests. Higher scores indicate better attention and executive function.
Changes of Trail Making Test scores from baseline to the end of 8 weeks | Baseline and 8 weeks
  Trail Making Test includes Part A(TMT-A) and Part B(TMT-B), that respectively evaluates attention and executive function via measuring the time in seconds required for completion of each part of the test. Higher scores indicate worse attention and executive function.
Changes of Rey Auditory Verbal Learning Test scores from baseline to the end of 8 weeks | Baseline and 8 weeks
  Rey Auditory Verbal Learning Test evaluates different aspects of verbal memory through measuring total learning, repetitions, delayed recall, retroactive interference, and proactive interference. Higher scores for total learning and delayed recall indicate better memory, while higher scores for repetitions, retroactive interference, and proactive interference indicate worse memory.
Changes of Stroop Test scores from baseline to the end of 8 weeks | Baseline and 8 weeks
  Stroop test consists of Stroop word test(Part A), Stroop color test(Part B) and Stroop color word test(Part C), that assess executive function through measuring the time in second required to complete each part and the number of errors for each part. Higher score for each part indicates worse executive function.
Changes of Rey-Osterrieth Complex Figure Test scores from baseline to the end of 8 weeks | Baseline and 8 weeks
  Rey-Osterrieth Complex Figure Test evaluates visuospatial construction ability through measuring the accuracy of copy, and evaluates visual memory via measuring the accuracies of immediate and delayed recalls. Higher scores indicate better visuospatial construction and visual memory.
Change of Verbal Fluency Test Scores from baseline to the end of 8 weeks. | Baseline and 8 weeks
  Verbal Fluency Test includes Phonemic Fluency Test, Category Fluency Test and Action Fluency Test, that evaluate language. Verbal Fluency Test measures the number of correct words produced under restricted search conditions of phonemic(letter F), category(animals) and action(kitchen actions). Higher score for each subtest indicates better language.
Change of Boston Naming Test from baseline to the end of 8 weeks | Baseline and 8 weeks
  Boston Naming Test includes 30 items and evaluates language through measuring the total of correct responses. The minimum score is 0, and the maximum score is 30. Higher score indicates better language.
Change of Multidimensional Fatigue Inventory score from baseline to the end of 8 weeks | Baseline and 8 weeks
  Multidimensional Fatigue Inventory is a self-report instrument consisting of 20-item devised to evaluate fatigue through measuring the dimensions of General Fatigue, Physical Fatigue, Mental Fatigue, Reduced Motivation and Reduced Activity. The minimum score is 20 ,and the maximum score is 100. Higher score indicate greater severity of fatigue.
Change of Pittsburgh Sleep Quality Index from baseline to the end of 8 weeks | Baseline and 8 weeks
  Pittsburgh Sleep Quality Index is a self-report questionnaire with 19 items, that assesses general sleep quality within 1 month through measuring the components of Subjective Sleep Quality, Sleep Latency, Sleep Duration, Habitual Sleep Efficiency, Sleep Disturbances, Use of Sleeping Medication, and Daytime Dysfunction. The total score ranges from 0 to 21. Higher score indicates worse sleep quality.
Change of the Generalized Anxiety Disorde-7 score from baseline to the end of 8 weeks | Baseline and 8 weeks
  Generalized Anxiety Disorde-7 is a self-report questionnaire with 7 items, that assesses the level of anxiety in the past two week. The minimum score is 0, and the maximum score is 21. Higher score indicates greater severity of anxiety.
Change of Hamilton Depression Scale from baseline to the end of 8 weeks | Baseline and 8 weeks
  Hamilton Depression Scale is the most commonly used instrument for the assessment of depression in clinical practice. It includes 24 items and assesses the level of depression through measuring factors of Anxiety/Somatization, Weight, Cognitive Impairment, Diurnal Variation, Retardation, Sleep Disturbance, and Hopelessness. The total score range is 0 to 76. Higher total score indicates greater level of depression.
Change of the MOS Item Short From Health Survey from baseline to the end of 8 weeks | Baseline and 8 weeks
  The MOS Item Short From Health Survey is a self-report instrument with 36 items, that assesses quality of life through measuring subscales of Physical Function, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health. Higher subscores indicate better quality of life.
The change in level of N-acetylaspartate(NAA)at each hippocampus from baseline to the end of 8 weeks. | Baseline and 8 weeks.
  The level of NAA will be represented as the NAA to total creatine (Cr) ratio which is measured by Proton Magnetic Resonance Spectroscopy(MRS).
The change in level of choline(Cho)at each hippocampus from baseline to the end of 8 weeks. | Baseline and 8 weeks
  The level of Cho will be represented as the Cho to total creatine (Cr) ratio which is measured by Proton Magnetic Resonance Spectroscopy(MRS)
The change in level of glutamate (Glu) at each hippocampus from baseline to the end of 8 weeks. | Baseline and 8 weeks
  The level of Glu will be represented as the Glu to total creatine (Cr) ratio which is measured by Proton Magnetic Resonance Spectroscopy(MRS)
The change in level of glutamine (Gln) at each hippocampus from baseline to the end of 8 weeks. | Baseline and 8 weeks
  The level of Gln will be represented as the Gln to total creatine (Cr) ratio which is measured by Proton Magnetic Resonance Spectroscopy(MRS)
The change in level of lactate (Lac) at each hippocampus from baseline to the end of 8 weeks. | Baseline and 8 weeks
  The level of Lac will be represented as the Lac to total creatine (Cr) ratio which is measured by Proton Magnetic Resonance Spectroscopy(MRS)
The change in level of myo-inositol (mI) at each hippocampus from baseline to the end of 8 weeks. | Baseline and 8 weeks
  The level of mI will be represented as the mI to total creatine (Cr) ratio which is measured by Proton Magnetic Resonance Spectroscopy(MRS)
The change in level of glycerophosphorylcholine (GPC) at each hippocampus from baseline to the end of 8 weeks. | Baseline and 8 weeks
  The level of GPC will be represented as the GPC to total creatine (Cr) ratio which is measured by Proton Magnetic Resonance Spectroscopy(MRS)
The change in level of glutathione (GSH) at each hippocampus from baseline to the end of 8 weeks. | Baseline and 8 weeks
  The level of GSH will be represented as the GSH to total creatine (Cr) ratio which is measured by Proton Magnetic Resonance Spectroscopy(MRS)
The change of resting-state functional connectivity(RSFC) at each hippocampus from baseline to the end of 8 weeks. | Baseline and 8 weeks
  The RSFC for each hippocampus will be examined with functional Magnetic Resonance Imaging(fMRI).

OTHER OUTCOMES:
The number of participants with treatment-related adverse events recorded in Case Report Form(CRF) at the end of treatment at 8 weeks | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided
There is not a plan to make individual participant data (IPD) available to other researchers at this time.